CLINICAL TRIAL: NCT00001746
Title: Evaluation of Patients With Known or Suspected Inherited Heart Disease (Screening Protocol)
Brief Title: Screening for Inherited Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980102; 98-H-0102
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2003-04

CONDITIONS: Heart Disease; Hypertrophic Cardiomyopathy
Keywords: Hypertrophic Cardiomyopathy; HCM; Evaluation for Research; Medical Advice
MeSH Terms: conditions — Heart Diseases; Cardiomyopathy, Hypertrophic

SUMMARY:
Genetically inherited heart diseases like hypertrophic cardiomyopathy (HCM) are conditions affecting the heart passed on to family members by abnormalities in genetic information. These conditions are responsible for many heart related deaths and illnesses.

Presently, there are several research studies being conducted in order to improve the understanding of disease processes and symptoms associated with genetically inherited heart diseases.

This study is designed to determine the eligibility of patients diagnosed with or suspected to have inherited heart disease to participate in these research studies.

DETAILED DESCRIPTION:
Patients with hypertrophic cardiomyopathy (HCM) and other inherited cardiac diseases are being studied under several research protocols to determine their pathogenesis and clinical manifestations. The purpose of this protocol is to determine the eligibility of patients with known or suspected inherited heart conditions for our research protocols.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects and family members known or suspected to have inherited a cardiac disease such as HCM.

EXCLUSION CRITERIA

Patients with cardiac conditions that are not known to be inherited.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-04; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Maron BJ, Bonow RO, Cannon RO 3rd, Leon MB, Epstein SE. Hypertrophic cardiomyopathy. Interrelations of clinical manifestations, pathophysiology, and therapy (1). N Engl J Med. 1987 Mar 26;316(13):780-9. doi: 10.1056/NEJM198703263161305. No abstract available. PMID 3547130
- [Background] Wigle ED, Rakowski H, Kimball BP, Williams WG. Hypertrophic cardiomyopathy. Clinical spectrum and treatment. Circulation. 1995 Oct 1;92(7):1680-92. doi: 10.1161/01.cir.92.7.1680. PMID 7671349
- [Background] Solomon SD, Jarcho JA, McKenna W, Geisterfer-Lowrance A, Germain R, Salerni R, Seidman JG, Seidman CE. Familial hypertrophic cardiomyopathy is a genetically heterogeneous disease. J Clin Invest. 1990 Sep;86(3):993-9. doi: 10.1172/JCI114802. PMID 1975599